## **Informed consent form**

## **Project title:**

Dispatcher-Assisted Cardiopulmonary Resuscitation: A Randomised Controlled Trial of Low-Dose, High-Frequency Simulation-Based Training and the Impact on Real Out-of-Hospital Cardiac Arrest Calls.

## Declaration from a participant in the research project:

I have been given written information, and I know enough about the project to say yes to participate.

I know that participating is voluntary and that I, at any point, can withdraw my consent.

I voluntarily consent to participate in the research and have been given a copy of the written information about the project for my use.

| Test subject name (capital letters): | |
|---|---|
| Date: Signature: | |
| Do you wish to be informed about the results of the research project? | |
| Yes (mark with x) No | (mark with x) |
| Declaration by the provider of information: | |
| I declare that the participant in the research project has been given written information about the project. | |
| In my opinion, sufficient information has been provided to enable participants to decide whether to participate or not. | |
| Name of the person who provided information: | |
| Date: Signature: | |

